CLINICAL TRIAL: NCT05447663
Title: A Phase Ib/II, Open Label Study of Siremadlin Monotherapy and in Combination With Donor Lymphocyte Infusion as a Treatment for Patients With Acute Myeloid Leukemia Post-allogeneic Stem Cell Transplantation Who Are in Complete Remission But at High Risk for Relapse.
Brief Title: A Study of Siremadlin Alone and in Combination With Donor Lymphocyte Infusion in Acute Myeloid Leukemia Post-allogeneic Stem Cell Transplant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study has been stopped following the strategic decision from the Sponsor. Not based on any safety findings or safety concerns with siremadlin.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHDM201K12201; 2021-003596-34 (EudraCT Number)
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; Allogeneic Stem Cell Transplantation
Keywords: Acute Myeloid Leukemia; Acute myeloid leukemia post allogeneic stem cell transplantation; AML; allogeneic stem cell transplantation; HDM201; siremadlin; donor lymphocyte infusion; DLI; MDM2; p53; allo-SCT
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — siremadlin

STUDY DESIGN:
Intervention Model Description: Study started out a phase l/ll study but because it was terminated, it never made it to phase ll.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Siremadlin (HDM201) (Experimental): Participants with AML post allogeneic stem cell transplantation (allo-SCT) received siremadlin monotherapy in part 1 and were to have received siremadlin monotherapy as well as in combination with donor lymphocyte infusion in part 2.
  Interventions: Drug: Siremadlin

INTERVENTIONS:
Drug: Siremadlin — Siremadlin was administered at a starting dose of 30 mg/day on days 1-5 of a 28-day treatment cycle (Part 1).
  Other Names: HDM201

SUMMARY:
The purpose of this study was to confirm a safe dose and schedule as well as the preliminary efficacy of siremadlin alone, and in combination with donor lymphocyte infusion (DLI), in adult participants with Acute Myeloid Leukemia (AML) who were in remission following allogeneic stem cell transplantation (allo-SCT) but were at high risk for relapse based on the presence of pre-transplant risk factors.

DETAILED DESCRIPTION:
This is a Phase Ib/II, single arm, open label, multi-center study of siremadlin as monotherapy and in combination with DLI, in adult participants with AML.

The primary purpose of the study was to confirm the safe dose and schedule of siremadlin monotherapy and in combination with DLI. The study is also designed to assess the preliminary efficacy in preventing hematologic relapse.

The study was initially planned to enroll approximately 38 participants starting with a dose confirmation of siremadlin monotherapy (part 1) to determine the siremadlin recommended dose, followed by a treatment strategy of siremadlin/DLI (Part 2).

After enrolling 8 participants (at the starting dose 30 mg/day on days 1-5 of a 28-day treatment cycle) in part 1, Novartis took the decision to put the enrollment in permanent halt and terminate the siremadlin program. For that reason, the enrollment in part 2 will not be open. The Novartis decision was not driven by any safety concerns.

In part 1 approximately 12 participants were planned to be enrolled in 2 cohorts (starting dose 30 mg/day on days 1-5 of a 28-day treatment cycle, dose level +1 at 40 mg/day and dose level -1 at 20 mg/day) and participants were planned to be treated for a maximum of 24 cycles.

In part 2, participants were planned to follow a treatment strategy, which contains three consecutive phases for a maximum of 24 cycles in total:

* A priming phase with siremadlin monotherapy at the recommended dose determined in Part 1 (for at least 2 cycles). Participants who were not eligible for the combination phase of siremadlin/DLI could continue priming phase with siremadlin monotherapy.
* A combination phase of siremadlin in combination with DLI (siremadlin/DLI) for participants who were eligible to receive DLI (up to a total of 3 combination cycles).
* A maintenance phase with siremadlin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with AML diagnosis, who underwent one allo-SCT to treat AML and are currently at ≥ Day 60 but no later than Day 120 (≤ Day 120) post allo-SCT.
* Pre-allo-SCT - Participants must have any of the following risk factors that put them at high risk for relapse:

  • AML in first CR (CR1) prior to allo-SCT with one of the following:
* Adverse risk genetic abnormalities per 2017 ELN risk stratification. Patients with TP53 mutant AML at diagnosis are eligible if they meet eligibility criteria.
* Therapy-related AML (t-AML).
* Secondary AML (sAML) [AML secondary to antecedent myelodysplastic syndrome (MDS) or AML secondary to myeloproliferative neoplasm (MPN)].

  • AML in second or greater CR (≥CR2) prior to allo-SCT.
* Allo-SCT must have the following characteristics:

  * Unmanipulated/T cell-replete bone marrow or peripheral blood stem cells as a graft source.
  * Matched related (family) donor (MFD) or matched unrelated donor (MUD): Human Leukocyte Antigen (HLA) matching of donor and recipient should be at a minimum of 8/8 antigen or allele matched at HLA-A, -B, -C, -DRB1 loci.
  * Any conditioning regimen intensity is permitted, the use of anti-thymocyte globulin (ATG) or alemtuzumab or post-transplant cyclophosphamide as a part of conditioning is allowed.
* Donor lymphocytes are collected, cryopreserved and available for infusion (DLI), or obtaining donor lymphocytes for DLI is feasible (applicable only for part 2)
* Post-allo-SCT, participants must have achieved CR or CRi with no current evidence of hematologic relapse
* Eastern Cooperative Oncology Group (ECOG ) performance status 0, 1 or 2.
* Laboratory test results indicating adequate liver and kidney function laboratory test results
* Evidence of adequate engraftment: Absolute Neutrophil Count (ANC) ≥ 1.0x109/L, Platelets (PLT) ≥ 75x109/L, Hemoglobin (Hgb) ≥ 8 g/dL (within 14 days prior to start of study treatment)

Exclusion criteria:

* Prior exposure to MDM-inhibitor
* Active acute GvHD (aGvHD) of any grade (per Harris et al 2016) and/or active chronic GvHD (cGvHD ) of any grade (per NIH criteria (Jagasia et al 2015)) requiring systemic therapy at time of study treatment initiation
* Past history of grade III or IV aGvHD and/or past history of moderate or severe cGvHD. History of lower grades of GvHD is permitted if GvHD resolved to grade 0 for at least 4 weeks prior to start of study treatment.
* Recipient of allo-SCT from MUD with ≥1 antigen or allele mismatch at HLA-A, -B, -C, -DRB1 locus (HLA matching < 8/8 antigens)
* Recipient of allo-SCT from a haploidentical family donor; and recipients of cord blood transplant as a graft source
* Prior systemic AML-directed treatments given at any time after allo-SCT (including DLI)
* Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half-lives or 4 weeks prior to starting study, whichever is longer
* GI disorders that may prevent the intake and absorption of oral siremadlin (eg, diarrhea, uncontrolled nausea/vomiting, GI bleeding, etc).
* Any concurrent severe and/or active uncontrolled bacterial, viral or fungal infection requiring parenteral antibacterial, antiviral or antifungal therapy. Prophylactic antimicrobial use (oral or parenteral) is allowed.
* Participants who require treatment with moderate or strong CYP3A inducers within 14 days prior to starting study treatment, or are expected to receive moderate or strong CYP3A inducers during the entire study
* Cardiac or cardiac repolarization abnormality, that are clinically significant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Germany (2):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Freiburg im Breisgau
- Italy (2):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 participants were planned to be enrolled; 12 participants in Part 1 and 26 participants in Part 2; however, due to permanent recruitment halt, the enrollment was stopped after the 1st dose escalation meeting. The study was conducted in 6 centers in 3 countries: Germany, Italy and Spain.
Pre-assignment Details: Prior to dosing at Cycle 1 Day 1, participants who fulfilled all the inclusion/exclusion criteria were enrolled via IRT and a treatment number was provided for the study treatment siremadlin.
Groups:
- Siremadlin (HDM201) 30mg: Participants with AML post allogeneic stem cell transplantation (allo-SCT) received 30mg siremadlin monotherapy
Period: Overall Study
Arm/Group | Siremadlin (HDM201) 30mg
Started | 8
Entered Post-treatment Follow-up | 7
Did Not Enter Post-treatment Follow-up | 1
On 10mg (Due to Concomitant Medication to Prevent Overexposure) | 1
Completed (Not completed = Discontinued from study, not treatment) | 0
Not Completed | 8
Not completed — Study terminated by Sponsor | 5
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): FAS comprises all participants who received any study drug (i.e., at least one dose of siremadlin with or without Donor lymphocyte infusion (DLI)). Only the siremadlin 30 mg arm was opened for enrollment in the study.
Arm/Group | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (17.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 7
  Hispanic or Latino | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Dose Limiting Toxicities (DLTs) With Siremadlin Monotherapy in Part 1 (Dose Confirmation With Siremadlin Monotherapy)
Description: To determine the dose and schedule of siremadlin monotherapy that are tolerable without unacceptable toxicities as defined by the incidence of DLT during the first cycle of treatment in part 1. 'A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed, by the Investigator, to be at least possibly related to study treatment (siremadlin monotherapy and/or siremadlin in combination with Donor lymphocyte infusion (DLI)), and as unrelated to disease, disease progression, inter-current illness, or concomitant medications, that occurs during the DLT observation period and meets severity criteria as per protocol.
Time Frame: from cycle 1 day 1 (C1D1) to end of Cycle 1 (cycle = 28days)
Population: Dose Determining Set (DDS): The Dose Determining Set (DDS) includes participants in the dose determination phase who met specific treatment cycles, exposure criteria, follow-up/DLT observation, and safety evaluations, or experienced a DLT during the observation period. Only the 30 mg siremadlin arm was opened for enrollment, and patients needing dose reduction during Cycle 1 were not analyzed separately.
Measure: Count of Participants; unit: Participants
Groups:
- Siremadlin (HDM201) 30mg: Participants with AML post allogeneic stem cell transplantation (allo-SCT) received 30mg siremadlin monotherapy in part 1
Arm/Group | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 7
Participants | 1

2. Primary Outcome: Time to Dose Limiting Toxicity (DLT) With Siremadlin in Combination With Donor Lymphocyte Infusion (DLI), in Part 2
Description: To determine the dose and schedule of siremadlin in combination with DLI that are tolerable without unacceptable toxicities (siremadlin recommended dose for combination), defined as time from start of combination phase to first DLT observed during the entire combination phase.
Time Frame: From Day 1 of combination Cycle 1 to Day 42 of the last cycle of combination phase (up to 3 cycles of siremadlin/DLI combination). Cycle duration: 42 days
Population: Part 2 did not open for enrollment due to recruitment halt, so no data was analyzed hence no data to report.
Groups:
- Siremadlin (HDM201) + DLI: Participants with AML post allogeneic stem cell transplantation (allo-SCT) who were to have received siremadlin in combination with Donor Lymphocytes Infusion (DLI) in part 2
Arm/Group | Siremadlin (HDM201) + DLI
Number analyzed (Participants) | 0

3. Primary Outcome: Percentage of Participants Who Are Alive and Maintained Complete Remission (CR) or Complete Response With Incomplete Hematological Recovery (CRi) With no Evidence of Hematologic Relapse (Part 2)
Description: This involves evaluating the preliminary efficacy of siremadlin (as monotherapy, in priming and/or maintenance, with or without siremadlin in combination with DLI) on the prevention of hematologic relapse.
Time Frame: Over 6 months from start of study treatment strategy (part 2 - siremadlin/DLI treatment strategy)
Population: Part 2 did not open for enrollment due to recruitment halt, so no data was analyzed hence no data to report.
Arm/Group | Siremadlin (HDM201) + DLI
Number analyzed (Participants) | 0

4. Secondary Outcome: Participants Who Are Alive and Maintained CR or CRi With no Evidence of Hematologic Relapse (Part 1 -Siremadlin Monotherapy at the Recommended Dose for Part 2 )
Description: This involves evaluating the preliminary efficacy of siremadlin monotherapy at the recommended dose for part 2 on prevention of hematologic relapse
Time Frame: Over 6 months from start of siremadlin monotherapy (part 1)
Population: Participants who received siremadlin monotherapy at the recommended dose for Part 2. The recommended dose for Part 2 could not be determined and therefore there were no patients meeting the reporting criteria for this endpoint.
Arm/Group | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Time From Start of Study Treatment to the Date of First Documented Hematologic Relapse or Death Due to Any Cause, Whichever Occurs First
Description: Assessment of relapse free survival (RFS) in part 2
Time Frame: From start of study treatment to up to 36 months from last patient first treatment
Population: Part 2 did not open for enrollment due to recruitment halt, so no data was analyzed hence no data to report.
Arm/Group | Siremadlin (HDM201) + DLI
Number analyzed (Participants) | 0

6. Secondary Outcome: Cumulative Incidence of AML Relapse at 1 Year and 2 Years After Start of Study Treatment
Description: Cumulative incidence of Acute Myeloid Leukemia (AML) relapse at one year and 2 years after the start of study treatment in part 1 and 2. Cumulative incidence of relapse (CIR) is defined as the time from start of study treatment to the date of first documented hematologic relapse. CIR was to be analyzed in the FAS population who initiated priming phase at siremadlin recommended dose (RD) in Part 2 and participants at the RD in Part 1.
Time Frame: 1 year and 2 years after start of study treatment
Population: Participants who received siremadlin at the recommended dose (RD) for Part 2 and had available efficacy data at 1 year and 2 years after start of study treatment. The RD for Part 2 could not be determined and there were no patients with efficacy data collected at 1 year and 2 years after start of study treatment. Therefore, there were no patients meeting the reporting criteria for this endpoint.
Arm/Group | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 0

7. Secondary Outcome: Time From Start of Study Treatment to the Date of Death From Any Cause
Description: Assessment of Overall survival (OS) in part 2
Time Frame: From start of study treatment to up to 36 months from last patient first treatment
Population: Part 2 did not open for enrollment due to recruitment halt, so no data was analyzed hence no data to report.
Arm/Group | Siremadlin (HDM201) + DLI
Number analyzed (Participants) | 0

8. Secondary Outcome: Incidence of Graft Versus Host Disease (GvHD)
Description: Incidence of grade III or IV acute GvHD, and moderate to severe chronic GvHD in part 1. Part 2 never started.
Time Frame: From start of study treatment up to approx. 8 months
Population: Safety Set: Safety set includes all participants from the Full Analysis Set (FAS), i.e. all participants who received any study drug (i.e., at least one dose of siremadlin with or without DLI). Only the siremadlin 30 mg arm was opened for enrollment, and patients requiring any dose reduction throughout the study were not analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 8
Participants
  Grade 3 acute GvHD | 2
  Moderate chronic GvHD | 1

9. Secondary Outcome: Percentage of Participants With Permanent Study Treatment Discontinuation Due to GvHD or Other Adverse Events
Description: Percentage of participants with permanent discontinuation of study treatment due to GvHD or other adverse events in part 1. As part 2 was not started, there were no participants to analyze in part 2.
Time Frame: From start of study treatment up to approx. 8 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 8
Participants | 3

10. Secondary Outcome: Time From Start of Study Treatment to the Date of First Documented Occurrence or Worsening of Treatment Emergent Grade III or IV Acute GvHD, or Chronic GvHD Requiring Initiation of Systemic Immunosuppressive Treatment
Description: Assessment of GvHD-free/relapse-free survival (GRPF) in Part 1 and 2. According to the study protocol, time-to-event endpoints in Part 1 were planned to be analyzed using Kaplan-Meier method only for participants who received siremadlin at the recommended dose for Part 2.
Time Frame: From start of treatment up to approx. 8 months
Population: Participants who received siremadlin monotherapy at the recommended dose for Part 2, and participants enrolled in Part 2. The recommended dose for Part 2 could not be determined and Part 2 was not opened, and therefore there were no patients meeting the reporting criteria for this endpoint.
Arm/Group | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Pharmacokinetic (PK) Characteristic AUC of Siremadlin
Description: AUC is the area under the concentration vs. time curve in part 1 and was based on plasma concentration. Part 2 did not open for enrollment due to recruitment halt and so no data was analyzed.
  AUClast: The AUC from time zero to the last quantifiable concentration point (Tlast) (mass x time x volume-1).
  AUC0-t: The area under the concentration vs. time Curve (AUC) from time zero to specified time point.
Time Frame: AUC from time 0 to 8hr postdose, AUC0- 8hr (Cycle 1 Day 1, Cycle 1 Day 5) in part 1 [each cycle is 28 days for monotherapy]
Population: Pharmacokinetic Analysis Set (PAS): PAS includes all participants in the safety set who provide at least one evaluable PK concentration of siremadlin. One participant from the 30mg cohort received a siremadlin reduced dose of 10 mg due to coadministration of a strong CYP3A4 inhibitor as per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Siremadlin (HDM201) 10mg: Participants with AML post allogeneic stem cell transplantation (allo-SCT) received 10mg siremadlin monotherapy
Arm/Group | Siremadlin (HDM201) 10mg | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 1 | 7
hr*ng/mL
  AUClast: Cycle 1 Day 1 | 1497 (NA) — NA: Data could not be analyzed as there was only 1 patient | 3077 (39.7)
  AUC0-8hr: Cycle 1 Day 1 | 446 (NA) — NA: Data could not be analyzed as there was only 1 patient | 1187.1 (39.8)
  AUClast: Cycle 1 Day 5: number analyzed (Participants) | 0 | 6
  AUClast: Cycle 1 Day 5 |  | 1880.7 (31.2)
  AUC0-8hr: Cycle 1 Day 5: number analyzed (Participants) | 0 | 6
  AUC0-8hr: Cycle 1 Day 5 |  | 1894 (30.3)

12. Secondary Outcome: PK Characteristic Cmax of Siremadlin
Description: The maximum (peak) observed plasma drug concentration following drug administration (mass x volume^-1) in part 1. Part 2 did not open for enrollment due to recruitment halt and so no data was analyzed.
Time Frame: from 0 to 24 hrs post-dose (Cycle 1 Day 1), from 0 to 8 hr post-dose (Cycle 1 Day 5) in part 1 [each cycle is 28 days for monotherapy]
Population: Pharmacokinetics Analysis Set (PAS): PAS includes all participants in the safety set who provide at least one evaluable PK concentration of siremadlin. One participant from the 30mg cohort received a siremadlin reduced dose of 10 mg due to coadministration of a strong CYP3A4 inhibitor as per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Siremadlin (HDM201) 10mg | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 1 | 7
ng/mL
  Cycle 1 Day 1 | 73.6 (NA) — NA: Data could not be analyzed as there was only 1 patient | 207.68 (36.2)
  Cycle 1 Day 5: number analyzed (Participants) | 0 | 6
  Cycle 1 Day 5 |  | 296.92 (30.4)

13. Secondary Outcome: PK Characteristic Tmax of Siremadlin
Description: The time to reach maximum (peak) plasma drug concentration after drug administration (time) in part 1. Part 2 did not open for enrollment due to recruitment halt and so no data was analyzed.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Siremadlin (HDM201) 10mg | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 1 | 7
hour (hr)
  Cycle 1 Day | 3.00 [3.00 to 3.00] | 5.95 [2.02 to 6.03]
  Cycle 1 Day 5: number analyzed (Participants) | 0 | 6
  Cycle 1 Day 5 |  | 4.50 [1.92 to 7.75]

14. Secondary Outcome: PK Characteristic Ctrough of Siremadlin
Description: Concentration that is just prior to the beginning of, or at the end of a dosing interval; corresponding to the pre-dose concentration in part 1 and 2. Part 2 never started.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 5 in part 1; [each cycle is 28 days]
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Siremadlin (HDM201) 10mg | Siremadlin (HDM201) 30mg
Number analyzed (Participants) | 1 | 7
ng/mL
  Cycle 1 Day 1 (Pre-dose) | 0 (0) | 0 (0)
  Cycle 1 Day 5 (Pre-dose): number analyzed (Participants) | 0 | 6
  Cycle 1 Day 5 (Pre-dose) |  | 146.77 (79.726)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to 30 days after last dose of study treatment (on-treatment). Subjects remaining in the study after end of treatment (EOT) (responders and non-responders, regardless of when treatment was discontinued) were followed up to approx. 8 months to collect long term data survival including: survival, relapse/progression of the underlying hematologic disease.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Only the siremadlin 30 mg arm was opened for enrollment, and patients requiring any dose reduction throughout the study were not analyzed separately.
Arm/Group | Siremadlin (HDM201) 30mg
All-Cause Mortality (participants affected / at risk) | 2/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Siremadlin (HDM201) 30mg (N=8)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Abdominal infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Siremadlin (HDM201) 30mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Tachycardia (Cardiac disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Corneal exfoliation (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Mucosal inflammation (General disorders) | 1
Pyrexia (General disorders) | 3
Acute graft versus host disease (Immune system disorders) | 2
Chronic graft versus host disease (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Weight decreased (Investigations) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Endometrial thickening (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT05447663/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT05447663/SAP_001.pdf